CLINICAL TRIAL: NCT03979664
Title: Efficacy of Dexamethasone Iontophoresis in Psoriasis
Brief Title: Iontophoresis in Psoriasis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: FDA did not provide approval of the use of the drug for the study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00058450
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Psoriasis; Psoriasis Vulgaris; Skin Diseases
Keywords: Skin Lesions
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Subjects who meet the selection criteria will be offered an opportunity to take part in this study. This will be a prospective controlled study. After written informed consent, 20 subjects with symmetric thick plaque psoriasis lesions on the extremities and/or trunk will be enrolled and randomized to receive one activated iontophoresis patch containing dexamethasone sodium phosphate and another inactive control iontophoresis patch containing dexamethasone sodium phosphate on each limb containing a thick psoriatic plaque. Members of the research team will apply the patches. After application of the patch, subjects will be asked to return to the clinic in 1 week and 2 weeks. Efficacy will be measured at the 1-week and 2-week follow-up visit using a scale for erythema, scale, and thickness called the static Physician Global Assessment (sPGA) and subject satisfaction to treatment will be measured at the 2 week-follow-up using the PsoSat Questionnaire.
Who Masked: Participant
Masking Description: Without the subject knowing, one patch will be turned on whereas the other patch will be turned off. The patch will be turned on pulling a tab found in the middle of the butterfly-shaped patch. The other patch will be turned off by not pulling the tab found in the middle of the butterfly-shaped patch.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Iontophoresis (Active Comparator): One active iontophoresis patch will be applied once at the baseline clinical visit. The iontophoresis patches are called Activapatch intellidose 2.5.
  Interventions: Device: Activapatch intellidose 2.5 using active Iontophoresis; Drug: Dexamethasone
- Inactive Iontophoresis (Sham Comparator): One inactive iontophoresis patch will be applied once at the baseline clinical visit. The iontophoresis patches are called Activapatch intellidose 2.5.
  Interventions: Device: Activapatch intellidose 2.5 using inactive Iontophoresis

INTERVENTIONS:
Device: Activapatch intellidose 2.5 using active Iontophoresis — Iontophoresis is a drug delivery system that uses electromigration and electro-osmosis to move charged molecules. Electromigration is the movement of ions across the skin by an electrical field. Positive ions move away from a cathode (positive charge) and towards an anode (negative charge). Negative ions move away from an anode and towards a cathode. Electro-osmosis is the volume movement of positive ions away from the opposite charge. Since skin is negatively charge, positively charged ions penetrate deep in the tissue from the negatively charged skin. 4 The use of iontophoresis was incorporated into medicine in efforts to increase the penetration of medications and avoid injection procedures. Dexamethasone sodium phosphate 4 mg/mL vial will be used in the study. Using a syringe, 2 cc of dexamethasone will be drawn and poured onto the designated medication site on the iontophoresis patch. Once the medication is poured, the patch will be applied on the skin and turned on.
  Arms: Active Iontophoresis
Device: Activapatch intellidose 2.5 using inactive Iontophoresis — Iontophoresis is a drug delivery system that uses electromigration and electro-osmosis to move charged molecules. Electromigration is the movement of ions across the skin by an electrical field. Positive ions move away from a cathode (positive charge) and towards an anode (negative charge). Negative ions move away from an anode and towards a cathode. Electro-osmosis is the volume movement of positive ions away from the opposite charge. Since skin is negatively charge, positively charged ions penetrate deep in the tissue from the negatively charged skin. 4 The use of iontophoresis was incorporated into medicine in efforts to increase the penetration of medications and avoid injection procedures. Inactive medication will be used in the study. Using a syringe, 2 cc of inactive medication will be drawn and poured onto the designated medication site on the iontophoresis patch. Once the medication is poured, the patch will be applied on the skin and turned on.
  Arms: Inactive Iontophoresis
Drug: Dexamethasone — Dexamethasone sodium phosphate 4 mg/mL vial will be used in the study. Using a syringe, 2 cc of dexamethasone will be drawn and poured onto the designated medication site on the iontophoresis patch. Once the medication is poured, the patch will be applied on the skin and turned on.
  Arms: Active Iontophoresis

SUMMARY:
Iontophoresis potentially may be a good alternative to improved delivery of corticosteroids. Study Investigators propose to use iontophoresis to increase dexamethasone delivery into thick psoriasis plaques. The primary purpose of this study is to assess whether dexamethasone sodium phosphate iontophoresis is an effective local therapy for psoriasis. The objective of the study is to determine the efficacy of dexamethasone sodium phosphate iontophoresis for psoriasis.

DETAILED DESCRIPTION:
Subjects who meet the selection criteria will be offered an opportunity to take part in this study. This will be a prospective controlled study. After written informed consent, 20 subjects with symmetric thick plaque psoriasis lesions on the extremities and/or trunk will be enrolled and randomized to receive one activated iontophoresis patch containing dexamethasone sodium phosphate and another inactive control iontophoresis patch containing dexamethasone sodium phosphate on each limb containing a thick psoriatic plaque. Members of the research team will apply the patches. After application of the patch, subjects will be asked to return to the clinic in 1 week and 2 weeks. Efficacy will be measured at the 1-week and 2-week follow-up visit using a scale for erythema, scale, and thickness called the static Physician Global Assessment (sPGA) and subject satisfaction to treatment will be measured at the 2 week-follow-up using the PsoSat Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age.
* Subjects with diagnosed plaque-type psoriasis that is stable.
* Similar psoriasis plaques found on each limb and/or different sides of the trunk.
* Willingness to attend all scheduled visits and complete the study.
* Ability to understand and sign an informed consent form.

Exclusion Criteria:

* Known allergy to dexamethasone or any component of the formulation and iontophoresis components.
* Change in the use of systemic therapy in psoriasis within 4 weeks prior to applying iontophoresis patches (to allow time for washout).
* Use of topical therapy (including coal tar, salicylic acid, topical corticosteroids, vitamin D, vitamin A, urea) or recent phototherapy for psoriasis within 2 weeks prior to applying iontophoresis patches (to allow time for washout).
* Pregnancy or breast feeding women.
* Any other condition, in the judgement of the investigator, would put the subject at unacceptable risk to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Static Physician Global Assessment baseline | Baseline
  Static Physician Global Assessment of severity integrates all lesions for overall score. This measure is commonly used as a quick way to quantify disease severity both for clinical studies and non-clinical studies. Scores range from 0=clear to 5=very severe disease. Lower scores denote better outcomes.
Static Physician Global Assessment Week 1 | Change from Baseline to Week 1
  Static Physician Global Assessment of severity integrates all lesions for overall score. This measure is commonly used as a quick way to quantify disease severity both for clinical studies and non-clinical studies. Scores range from 0=clear to 5=very severe disease. Lower scores denote better outcomes.
Static Physician Global Assessment Week 2 | Change from Week 1 to Week 2
  Static Physician Global Assessment of severity integrates all lesions for overall score. This measure is commonly used as a quick way to quantify disease severity both for clinical studies and non-clinical studies. Scores range from 0=clear to 5=very severe disease. Lower scores denote better outcomes.

SECONDARY OUTCOMES:
PsoSat Questionnaire | Measured at Week 2
  PsoSat Questionnaire measures patient satisfaction to treatment. This measure was validated. PsoSat Questionniare consists of 8 items that are measured on a 5-item Likert scale. 0= poor agreement to 4= perfect agreement. Higher scores denote better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Feldman, MD, Ph.D, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koo J. Population-based epidemiologic study of psoriasis with emphasis on quality of life assessment. Dermatol Clin. 1996 Jul;14(3):485-96. doi: 10.1016/s0733-8635(05)70376-4. PMID 8818558
- [Background] Gelfand JM, Weinstein R, Porter SB, Neimann AL, Berlin JA, Margolis DJ. Prevalence and treatment of psoriasis in the United Kingdom: a population-based study. Arch Dermatol. 2005 Dec;141(12):1537-41. doi: 10.1001/archderm.141.12.1537. PMID 16365254
- [Background] Kimball AB, Jacobson C, Weiss S, Vreeland MG, Wu Y. The psychosocial burden of psoriasis. Am J Clin Dermatol. 2005;6(6):383-92. doi: 10.2165/00128071-200506060-00005. PMID 16343026
- [Background] Roustit M, Blaise S, Cracowski JL. Trials and tribulations of skin iontophoresis in therapeutics. Br J Clin Pharmacol. 2014 Jan;77(1):63-71. doi: 10.1111/bcp.12128. PMID 23590287
- [Background] Stefanou A, Marshall N, Holdan W, Siddiqui A. A randomized study comparing corticosteroid injection to corticosteroid iontophoresis for lateral epicondylitis. J Hand Surg Am. 2012 Jan;37(1):104-9. doi: 10.1016/j.jhsa.2011.10.005. PMID 22196293
- [Background] Chow C, Simpson MJ, Luger TA, Chubb H, Ellis CN. Comparison of three methods for measuring psoriasis severity in clinical studies (Part 1 of 2): change during therapy in Psoriasis Area and Severity Index, Static Physician's Global Assessment and Lattice System Physician's Global Assessment. J Eur Acad Dermatol Venereol. 2015 Jul;29(7):1406-14. doi: 10.1111/jdv.13132. Epub 2015 Apr 27. PMID 25917315
- [Background] Radtke MA, Spehr C, Reich K, Rustenbach SJ, Feuerhahn J, Augustin M. Treatment Satisfaction in Psoriasis: Development and Use of the PsoSat Patient Questionnaire in a Cross-Sectional Study. Dermatology. 2016;232(3):334-43. doi: 10.1159/000444635. Epub 2016 Apr 14. PMID 27073875
- [Background] Zempsky WT, Sullivan J, Paulson DM, Hoath SB. Evaluation of a low-dose lidocaine iontophoresis system for topical anesthesia in adults and children: a randomized, controlled trial. Clin Ther. 2004 Jul;26(7):1110-9. doi: 10.1016/s0149-2918(04)90183-x. PMID 15336476
- [Background] Le QV, Howard A. Dexamethasone iontophoresis for the treatment of nail psoriasis. Australas J Dermatol. 2013 May;54(2):115-9. doi: 10.1111/ajd.12029. Epub 2013 Feb 21. PMID 23425157